CLINICAL TRIAL: NCT03365674
Title: Vibration Anesthesia for Pain Reduction During Trigger Point Injection to the Gastrocnemius
Brief Title: Vibration for Pain Reduction During Trigger Point Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Young Eun Moon, Medical Doctor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPI vibrator
Record Dates: First submitted 2017-12-03; First posted 2017-12-07 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Myofascial Pain Syndromes
Keywords: Myofascial Pain Syndromes, Gastrocnemius, Trigger points, Injections, Vibration
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration group (Experimental): Vibrator head was applied (100Hz) on the popliteal fossa, during the trigger point injection
  Interventions: Device: Vibration
- Placebo group (Placebo Comparator): In placebo group, vibrator head was applied with switch-off sate, during the trigger point injection
  Interventions: Device: Placebo vibration

INTERVENTIONS:
Device: Vibration — Vibration applied with vibrator switch-on state (100Hz)
  Arms: Vibration group
Device: Placebo vibration — Vibrator applied with switch-off state
  Arms: Placebo group

SUMMARY:
The aim of this study is to evaluate the effects of vibration anesthesia for reducing pain induced by trigger point injection of gastrocnemius.

Sixty patients were randomized into the vibration or placebo group. In vibration groups, vibrator head was applied (100Hz) on the popliteal fossa, during the trigger point injection. In placebo group, same vibrator head was applied with switch-off sate. Then, a visual analog scale to evaluate the pain of trigger point injection and a five-point Likert scale for patients satisfaction were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have the trigger point in the gastrocnemius and show referred pain.

Exclusion Criteria:

* Those with prior history of trigger point injection
* Those with taking anti-platelet agent
* Those with hemorrhage tendency
* Pregnancy
* Acute infection
* those who were unable to understand a visual analog scale (VAS) or a Likert scale

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | Immediately after trigger point injection (within 5 minute)
  100 mm visual analog scale for evaluating the pain of trigger point injection

SECONDARY OUTCOMES:
5 point Likert scale for participant satisfaction | Immediately after trigger point injection (within 5 minute)
  5 point Likert scale to answer "Are you satisfied with the vibration application for reducing the pain of trigger point injection?"
5 point Likert scale for repeated usage | Immediately after trigger point injection (within 5 minute)
  5 point Likert scale to answer "Will you use the vibration application again if the trigger point injection is repeated in the future?"

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hyun Kim, MD,PhD, Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Hospital, Bucheon, Bucheon-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Yoon SH, Rah UW, Sheen SS, Cho KH. Comparison of 3 needle sizes for trigger point injection in myofascial pain syndrome of upper- and middle-trapezius muscle: a randomized controlled trial. Arch Phys Med Rehabil. 2009 Aug;90(8):1332-9. doi: 10.1016/j.apmr.2009.01.028. PMID 19651267
- [Background] Mally P, Czyz CN, Chan NJ, Wulc AE. Vibration anesthesia for the reduction of pain with facial dermal filler injections. Aesthetic Plast Surg. 2014 Apr;38(2):413-8. doi: 10.1007/s00266-013-0264-4. Epub 2014 Jan 24. PMID 24464122
- [Background] Park KY, Lee Y, Hong JY, Chung WS, Kim MN, Kim BJ. Vibration Anesthesia for Pain Reduction During Intralesional Steroid Injection for Keloid Treatment. Dermatol Surg. 2017 May;43(5):724-727. doi: 10.1097/DSS.0000000000001040. PMID 28244902
- [Derived] Moon YE, Kim SH, Seok H, Lee SY. Efficacy of Topical Vibratory Stimulation for Reducing Pain During Trigger Point Injection to the Gastrocnemius: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2019 Sep;100(9):1607-1613. doi: 10.1016/j.apmr.2019.02.010. Epub 2019 Mar 27. PMID 30926293